CLINICAL TRIAL: NCT03631823
Title: Linking the Gut Microbiota to the Prognosis of Glioblastoma Multiforme
Brief Title: Gut Microbiota and Glioblastoma Multiforme Prognosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Jinsong Wu, Professor, Huashan Hospital
Other Study IDs: GBM2018-2020
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Gut Microbiota, Glioblastoma Multiforme, Microglia, Tumor Related Macrophagocyte, Prognosis
MeSH Terms: conditions — Glioblastoma | interventions — Drug Therapy; Temozolomide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — microbiota DNA are extracted from human feces.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Radio/Chemotherapy group: The participants in this group receive the concurren radio/chemotrherapy
  Interventions: Other: Chemotherapy with temozolomide or no chemotherapy
- Radio/ without chemotherapy group: The participants in this group receive the radiotherapy but without chemotrherapy
  Interventions: Other: Chemotherapy with temozolomide or no chemotherapy
- Healthy volunteer group: The volunteers for control group
  Interventions: Other: Chemotherapy with temozolomide or no chemotherapy

INTERVENTIONS:
Other: Chemotherapy with temozolomide or no chemotherapy — This study is just an observational study.

SUMMARY:
Glioma is the most common primary cancer of the central nervous system, and around 50% of patients present with the most aggressive form of the disease, glioblastoma. Conventional therapies, including surgery, radiotherapy, and pharmacotherapy (typically chemotherapy with temozolomide), have not resulted in major improvements in the survival outcomes with only a median survival of around 15 months.The main reason may be related to the highly immunosuppressive tumor microenvironment. In recent years, the microbiome has emerged as a key regulator of not only systemic immune regulation but brain circuitry, neuro-physiology and microglia development. We hypothesized that there is a link between the gut microbiota and the GBM development and evolution through the immune regulation cells (microglia and tumor related macrophagocyte) in the blood circulation to impact the prognosis( PFS and MST) of GBM patients.

DETAILED DESCRIPTION:
We divide the paticipants into three groups. (total number = 200 subjects)

1. Radio/Chemotherapy group - 80 subjects
2. Radio/ without chemotherapy group - 70 subjects
3. Healthy volunteer group - 50 subjects

After the collection of stools before operation and 3 months after the operaton, we will analyze the composition and distribution of gut microbiota, and compare the results of three experiment groups.Then we will followe up the patients and analyze the correlation between gut microbiota and prognosis of GBM.

ELIGIBILITY:
Inclusion Criteria:

The participants diagnosed with glioblastoma multiforme by immunohistochemistry and molecular (IDH1, 1p19q, TERT) diagnosis of WHO 2016 classification of Gliomas.

The healthy volunteers.

Exclusion Criteria:

1. No cancer or IBD (inflammatory bowel disease);
2. No history of abdominal surgery;
3. No medication related to gastrointestinal motility within 3 months;
4. No oral antibiotic treatments previous 1 month before neurosurgery operation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients enrolled from neurosurgery department of Huashan hospital and the Shandong provincial hospital affiliated to Shandong University; while the healthy volunteers come from the health examination center of huashan hospital and Shandong provincial hospital affiliated to Shandong University.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-08-10 (Estimated); Primary Completion 2019-08-10 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Pre-operative gut microbiota in molecular subtype glioblastoma mutiforme multiform | 12 months
  To analysis the distribution and components of gut microbiota before operation
The perturbation of gut microbiota by temozolomide chemotherapy | 15 months
  To investigate the change of components of gut microbiota induced by chemotherapy
Link the gut microbiota and prognosis of GBM | 20 months
  To explore the correlation between the gut micriobiota and the prognosis (PFS and MST) by bioinformatic big data process.

CONTACTS AND LOCATIONS:
Overall Officials: Jinsong Wu, Ph.D. & M.D, Study Chair — Huashan Hospital; Weifeng Shi, Ph.D., Principal Investigator — Taishan Medical Univiersity; Yingchao Liu, Ph.D. & M.D, Study Director — Shandong provincial hospirtal affiliated to Shandong University

IPD SHARING:
Plan to Share IPD: No